CLINICAL TRIAL: NCT00628043
Title: A Phase Ⅲ Randomized Double-Blind Placebo-Controlled Study of Epoetin Beta for the Treatment of Chemotherapy-Induced Anemia (CIA) in Cancer Patients
Brief Title: Clinical Study of Epoetin Beta to Chemotherapy-Induced Anemia (CIA) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical Co., Ltd., Chugai Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EPO316 JP
Record Dates: First submitted 2008-02-24; First posted 2008-03-04 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Anemia
Keywords: Cancer; patients; with; chemotherapy; induced; anemia
MeSH Terms: conditions — Anemia; Neoplasms | interventions — epoetin beta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- EPOCH (Experimental)
  Interventions: Drug: epoetin beta
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: epoetin beta — Subcutaneous administration of epoetin beta 36,000 IU once-weekly for 12 weeks
  Arms: EPOCH
Drug: placebo — Subcutaneous administration of placebo once-weekly for 12 weeks
  Arms: placebo

SUMMARY:
This is a study to investigate the clinical efficacy and safety of epoetin beta 36,000 IU compared with placebo when administrated subcutaneously (s.c.) once-weekly for 12 weeks to anemic patients with lung cancer or gynecologic cancer undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer or gynecologic cancer patients
* Undergoing platinum-based chemotherapy repeated for ≧ 2 cycles after erythropoietin (EPO) or placebo administration
* 8.0 g/dL ≦ hemoglobin concentration (Hb) ≦ 10.0 g/dL
* 20 - 79 years old
* Performance status: 0 - 2
* No iron deficiency anemia

Exclusion Criteria:

* Red blood cell transfusion within 4 weeks before treatment
* Erythropoietin therapy within 8 weeks before treatment

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The proportion of the subjects who receive red blood cell (RBC) transfusion and/or hemoglobin (Hb) concentration < 8.0 g/dL | 16 weeks

SECONDARY OUTCOMES:
Change in Hb | 16 weeks
Change in FACT- total Fatigue Subscale score (FSS) | 16 weeks
Requirement for RBC transfusion | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yoshito Suzuki, Study Chair — Chugai Pharmaceutical
Locations (6):
- Japan (6):
  - Chugoku/Shikoku Region, Chugoku/Shikoku
  - Chubu Region, Chūbu
  - Hokkaido/Tohoku Region, Hokkaido/Tohoku
  - Kanto/Koshinetsu Region, Kanto/Koshinetsu
  - Kinki/Hokuriku Region, Kinki/Hokuriku
  - Kyushu Region, Kyushu